CLINICAL TRIAL: NCT02624791
Title: Evaluating and Improving Functional Driving Vision of Patients With Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Cox, PhD, Professor, Department of Psychiatry and NB Sciences, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15920
Record Dates: First submitted 2013-12-30; First posted 2015-12-08 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Astigmatism
Keywords: astigmatism, contact lens, driving
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: participants and research assistant blind to hypothesis
Oversight: Data Monitoring Committee: No

ARMS (6):
- Lens sequence 1 (Experimental): No contact lenses; 1-DAY ACUVUE® MOIST contact lenses;
  1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses
  Interventions: Device: 1-DAY ACUVUE® MOIST contact lenses; Device: 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses; Other: No contact lenses
- Lens sequence 2 (Experimental): No contact lenses; 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses;
  1-DAY ACUVUE® MOIST contact lenses
  Interventions: Device: 1-DAY ACUVUE® MOIST contact lenses; Device: 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses; Other: No contact lenses
- Lens sequence 3 (Experimental): 1-DAY ACUVUE® MOIST contact lenses; No contact lenses;
  1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses
  Interventions: Device: 1-DAY ACUVUE® MOIST contact lenses; Device: 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses; Other: No contact lenses
- Lens sequence 4 (Experimental): 1-DAY ACUVUE® MOIST contact lenses;
  1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses; No contact lenses
  Interventions: Device: 1-DAY ACUVUE® MOIST contact lenses; Device: 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses; Other: No contact lenses
- Lens sequence 5 (Experimental): 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses;
  1-DAY ACUVUE® MOIST contact lenses; No contact lenses
  Interventions: Device: 1-DAY ACUVUE® MOIST contact lenses; Device: 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses; Other: No contact lenses
- Lens sequence 6 (Experimental): 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses; No contact lenses;
  1-DAY ACUVUE® MOIST contact lenses
  Interventions: Device: 1-DAY ACUVUE® MOIST contact lenses; Device: 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses; Other: No contact lenses

INTERVENTIONS:
Device: 1-DAY ACUVUE® MOIST contact lenses — spherical contact lenses worn during simulated driving tests
Device: 1-DAY ACUVUE® MOIST for ASTIGMATISM contact lenses — toric contact lenses worn during simulated driving tests
Other: No contact lenses — simulated driving tests

SUMMARY:
Small amounts of astigmatism are often uncorrected in contact lens wearers. The effect with respect to driving is unknown, but it could threaten safe operation of a motor vehicle, especially under conditions such as nighttime driving when visual abilities are highly challenged. This study measures driving-specific visual abilities and simulated driving performance in participants with astigmatism who either have or do not have their astigmatism corrected. The primary hypothesis is that at a tactical level, contact lenses correcting for astigmatism will result in safer driving performance overall. The secondary hypothesis is that at an operational level, contact lenses correcting for astigmatism will result in better driving-specific visual performance.

DETAILED DESCRIPTION:
Safe driving relies heavily on "good vision." Good vision while driving relates to multiple abilities, such as dynamic visual acuity, contrast sensitivity, management of glare and peripheral vision, etc. While spherical contact lenses address issues of correction of visual acuity as determined by forward static vision tests, if they do not provide visual acuity both immediately and smoothly with eye movement then vision can be compromised. Glare can be a problem as well when contact lenses are off center. Fluctuating vision as a result of lens movement on the eye could be especially problematic and frustrating for patients who have astigmatism. Furthermore, experiencing moments of blurred vision no matter how brief can be potentially hazardous while driving. The 1*DAY ACUVUE® MOIST for ASTIGMATISM contact lenses have a unique blink-activated stabilization system to prevent rotation of the lens on the eye, and may have significant visual advantages for drivers with astigmatism. These lenses provide continuous corrected acuity compared to non-ballasted contact lenses, and thus are potentially safer for driving. Contact comparison will consist of 1*DAY ACUVUE® MOIST (spherical control) versus 1*DAY ACUVUE® MOIST for ASTIGMATISM (the daily disposable astigmatism alternative).

The study will investigate the potential advantages of contact lenses specifically designed to correct for astigmatism, compared to similar correction with spherical contacts, for adult licensed drivers with astigmatism, employing a double-blind (subjects and research assistant blind to hypotheses), randomized, cross-over design (spherical, vs. astigmatism contacts). This will be a multi-stage study comprised of the following:

Preliminary study to determine the likelihood of detecting a significant difference between the standard spherical and astigmatism contacts in a full Randomize Clinical Trial (n=12; data and power analysis)

ELIGIBILITY:
Inclusion Criteria:

* Adult licensed drivers between the ages of 18-39, similar number of males and females will be studied who meet the following inclusion criteria:
* Bilateral corrected vision of 20/40 or better
* Bilateral astigmatism between 0.75 to 2.0 diopters, with spherical correction from -1 to -6
* No active eye infection
* No defective peripheral vision
* Do not have correction for bifocals
* Routinely wear contact lenses more than 4 times per week
* Routinely drive a car more than 4 times week
* Do not have a history of motion, sea or big screen (e.g. IMAX) sickness or experience persistent Simulation Adaptation Syndrome

Exclusion Criteria:

* Bilateral corrected vision of worse than 20/40
* No astigmatism
* Active eye infection
* Defective peripheral vision
* Wear bifocals
* Wears contact lenses less than 4 times per week
* Drives infrequently (less than 4 times per week)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cox, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Driving Safety Lab, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cox DJ, Banton T, Record S, Grabman JH, Hawkins RJ. Does correcting astigmatism with toric lenses improve driving performance? Optom Vis Sci. 2015 Apr;92(4):404-11. doi: 10.1097/OPX.0000000000000554. PMID 25946099

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens Sequence 1: None; Sphere; Toric
- Lens Sequence 2: None; Toric; Sphere
- Lens Sequence 3: Sphere; None; Toric
- Lens Sequence 4: Sphere; Toric; None
- Lens Sequence 5: Toric; None; Sphere
- Lens Sequence 6: Toric; Sphere; None
Period: Overall Study
Arm/Group | Lens Sequence 1 | Lens Sequence 2 | Lens Sequence 3 | Lens Sequence 4 | Lens Sequence 5 | Lens Sequence 6
Started | 2 | 1 | 2 | 2 | 2 | 2
Completed | 0 | 1 | 2 | 2 | 2 | 2
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 11 participants completed the operational tests 9 participants completed the tactical tests
Groups:
- Contact Lens Sequence: Order in which each participant received the 3 lens conditions
Arm/Group | Contact Lens Sequence
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (4.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Tactical Composite Score
Description: Z-score composite of tactical testing outcomes
Time Frame: 1 day laboratory study
Measure: Mean (Standard Deviation); unit: Z score
Groups:
- Contact Lens Rx: All study participants
Arm/Group | Contact Lens Rx
Number analyzed (Participants) | 9
Z score
  None | -1.73 (3.53)
  Sphere | 0.19 (2.62)
  Toric | 1.54 (1.75)

2. Secondary Outcome: Operational Composite Score
Description: Z-score composite of operational testing outcomes
Time Frame: 1 day laboratory study
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Contact Lens Rx
Number analyzed (Participants) | 11
Z score
  None | -2.77 (4.30)
  Sphere | 1.37 (2.37)
  Toric | 1.40 (2.65)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Participants were assessed for Simulation Adaptation Syndrome by using a rating scale after each of their 3 simulated driving periods.
Groups:
- Contact Lens Rx: None; Sphere; Toric
Arm/Group | Contact Lens Rx
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes